CLINICAL TRIAL: NCT03036163
Title: Open-label Prospective Noncomparative Study of Safety, Tolerability and Pharmacokinetics of PBTZ169 After Single and Multiple Fasting Oral Administration in Increasing Doses in Healthy Volunteers
Brief Title: Phase 1 Study of PBTZ169
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nearmedic Plus LLC (Industry)
Collaborators: OCT LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PBTZ169-Z00-C01-1
Record Dates: First submitted 2016-09-14; First posted 2017-01-30 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — macozinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1 (Experimental): 6 male healthy volunteers each of whom received once single oral dose of PBTZ169 - 40 mg (1 capsule)
  Interventions: Drug: PBTZ169 - 40 mg
- Cohort 2 (Experimental): 6 male healthy volunteers each of whom received once single oral dose of PBTZ169 - 80 mg (2 capsules)
  Interventions: Drug: PBTZ169 - 80 mg
- Cohort 3 (Experimental): 6 male healthy volunteers each of whom received once single oral dose of PBTZ169 - 160 mg (4 capsules)
  Interventions: Drug: PBTZ169 - 160 mg
- Cohort 4 (Experimental): 6 male healthy volunteers each of whom received once single oral dose of PBTZ169 - 320 mg (8 capsules)
  Interventions: Drug: PBTZ169 - 320 mg
- Cohort 5 (Experimental): 6 male healthy volunteers each of whom received once single oral dose of PBTZ169 - 640 mg (16 capsules)
  Interventions: Drug: PBTZ169 - 640 mg
- Cohort 6 (Experimental): 5 male healthy volunteers each of whom received once daily for 14 days 320 mg of PBTZ169 (8 capsules 40 mg)
  Interventions: Drug: PBTZ169 - 320 mg (multiple administration)
- Cohort 7 (Experimental): 5 male healthy volunteers each of whom received once daily for 14 days 640 mg of PBTZ169 (16 capsules 40 mg)
  Interventions: Drug: PBTZ169 - 640 mg (multiple administration)

INTERVENTIONS:
Drug: PBTZ169 - 40 mg — 40 mg of PBTZ169 (1 capsule) orally once in fasting state
  Other Names: PBTZ169
  Arms: Cohort 1
Drug: PBTZ169 - 80 mg — 80 mg of PBTZ169 (2 capsules 40 mg) orally once in fasting state
  Other Names: PBTZ169
  Arms: Cohort 2
Drug: PBTZ169 - 160 mg — 160 mg of PBTZ169 (4 capsules 40 mg) orally once in fasting state
  Other Names: PBTZ169
  Arms: Cohort 3
Drug: PBTZ169 - 320 mg — 320 mg of PBTZ169 (8 capsules 40 mg) orally once in fasting state
  Other Names: PBTZ169
  Arms: Cohort 4
Drug: PBTZ169 - 640 mg — 640 mg of PBTZ169 (16 capsules 40 mg) orally once in fasting state
  Other Names: PBTZ169
  Arms: Cohort 5
Drug: PBTZ169 - 320 mg (multiple administration) — 320 mg of PBTZ169 (8 capsules 40 mg) orally once per day in fasting state for 14 days
  Other Names: PBTZ169
  Arms: Cohort 6
Drug: PBTZ169 - 640 mg (multiple administration) — 640 mg of PBTZ169 (16 capsules 40 mg) orally once per day in fasting state for 14 days
  Other Names: PBTZ169
  Arms: Cohort 7

SUMMARY:
Open-label prospective non-comparative safety, tolerability and pharmacokinetics ascending dose randomized cohort study of PBTZ169 (capsules 40 mg) in fasted healthy volunteers after single and multiple oral administration

DETAILED DESCRIPTION:
Open-label prospective non-comparative safety, tolerability and pharmacokinetics ascending dose randomized cohort study of PBTZ169 (capsules 40 mg) in adult man healthy volunteers after single and multiple oral fasting administration. Study was conducted in one study center in Russian Federation. The study included two stages:

* Stage 1 - single oral fasting administration with dose escalation in 5 cohorts 6 healthy man volunteers each in main groups (plus 1 back-up volunteer in every group);
* Stage 2 - multiple oral fasting administration with dose escalation in 2 cohorts 6 healthy man volunteers each in main groups (plus 1 back-up volunteer in every group).

Screening procedures for each cohort performed within 7 days before the drug prescription and after the end of administration period in previous cohort. Screening in cohorts 2 and 6 was started only after safety tolerability and PK data analysis of previous cohorts.

All volunteers met the study inclusion/exclusion criteria was included successively into the following cohorts on Stage 1 (actual data):

* Cohort 1 (C1) - 6 volunteers of the main group each of whom received once single dose of the drug - 1 capsule containing 40 mg of PBTZ169;
* Cohort 2 (C2) - 6 volunteers of the main group each of whom received once 80 mg of PBTZ169 (2 capsules 40 mg);
* Cohort 3 (C3) - 6 volunteers of the main group each of whom received once 160 mg of PBTZ169 (4 capsules 40 mg);
* Cohort 4 (C4) - 6 volunteers of the main group each of whom received once 320 mg of PBTZ169 (8 capsules 40 mg);
* Cohort 5 (C5) - 6 volunteers of the main group each of whom received once 640 mg of PBTZ169 (16 capsules 40 mg).

On Stage 2 (actual data):

* Cohort 6 (C6) - 5 volunteers of the main group each of whom received 320 mg of PBTZ169 (8 capsules 40 mg) once daily for 14 days;
* Cohort 7 (C7) - 5 volunteers of the main group each of whom received 640 mg of PBTZ169 (16 capsules 40 mg) once daily for 14 days.

Safety was assessed throughout the study. For every volunteer series of urine and venous blood samples was collected for the safety, tolerability and PK assessment of PBTZ169.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent received from a volunteer.
2. Man aged 18 to 45 years old, inclusive.
3. Body mass index of 18.5-25 kg/m2.
4. Verified diagnosis: "healthy" according to data of standard clinical, laboratory and instrumental examination methods performed at screening:

   * Absence of deviations of physical examination parameters and vital signs (systolic blood pressure - 100-129 mm Hg, inclusive; diastolic blood pressure - 70-89 mm Hg, inclusive; heart rate - 60-80 bpm, inclusive);
   * Absence of deviations of laboratory parameters (complete blood count, blood biochemistry, urinalysis and tests for HIV, HBV, HCV, syphilis);
   * Normal parameters of 12-lead ECG;
   * Normal results of photofluorographic or X-ray examination (the results received maximum 6 months before screening can be used).
5. Ability, according to investigators opinion, to comply with all requirements of the protocol.
6. Agreement to use double contraception method during the study participation and for 3 months after the test drug administration - combination of male condom with not less than one of the following methods:

   * female partner using hormonal contraception;
   * using aerosols, creams, suppositories and other agents containing spermicides;
   * female partner using intrauterine device

Exclusion Criteria:

1. Aggravated allergic history, including presence of at least one episode of drug allergy.
2. Chronic diseases of cardiovascular, bronchopulmonary, neuroendocrine systems, ENT and gastrointestinal, hepatic, renal, blood and cutaneous diseases.
3. Chronic diseases of eyes except for mild to moderate myopia, hypermetropia and astigmatism.
4. Gastrointestinal surgeries (except for appendectomy performed not less than 1 year before screening).
5. Acute infections within less than 4 weeks before screening.
6. Regular drug administration within less than 4 weeks before screening.
7. Regular administration or application (including topical) of hormonal drugs for more than 1 week within less than 45 days before the screening.
8. Administration of drugs exerting evident effects on hemodynamics, hepatic function, etc. (barbiturates, omeprazole, cimetidine, etc.) within less than 45 days before the screening.
9. Positive tests for narcotic and psychotropic agents.
10. Donation (450 mL of blood or plasma) within less than 3 months before the screening.
11. Intake of more than 10 U of alcohol per week (1 unit of alcohol is equivalent to 500 mL of beer, 200 mL of vine or 50 mL of strong alcoholic drink) or historical data on alcoholism, narcomania, drug abuse.
12. Mental illnesses.
13. Smoking within half a year before the screening.
14. Previous participation in this clinical study and withdrawal from it due to any reason.
15. Participation in other clinical studies of drugs within less than 6 months before the screening.
16. Planned conception or sperm donation during the study after the test drug administration or during 3 months after the date of drug administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 6 healthy volunteers each of whom received one single oral dose of PBTZ169 - 40 mg (1 capsule)
  PBTZ169 - 40 mg: 40 mg of PBTZ169 (1 capsule) orally once in fasting state
- Cohort 2: 6 healthy volunteers each of whom received one single oral dose of PBTZ169 - 80 mg (2 capsules)
  PBTZ169 - 80 mg: 80 mg of PBTZ169 (2 capsules 40 mg) orally once in fasting state
- Cohort 3: 6 healthy volunteers each of whom received one single oral dose of PBTZ169 - 160 mg (4 capsules)
  PBTZ169 - 160 mg: 160 mg of PBTZ169 (4 capsules 40 mg) orally once in fasting state
- Cohort 4: 6 healthy volunteers each of whom received one single oral dose of PBTZ169 - 320 mg (8 capsules)
  PBTZ169 - 320 mg: 320 mg of PBTZ169 (8 capsules 40 mg) orally once in fasting state
- Cohort 5: 6 healthy volunteers each of whom received one single oral dose of PBTZ169 - 640 mg (16 capsules)
  PBTZ169 - 640 mg: 640 mg of PBTZ169 (16 capsules 40 mg) orally once in fasting state
- Cohort 6: 5 healthy volunteers each of whom received а daily dose of 320 mg of PBTZ169 (8 capsules 40 mg) for 14 days
  PBTZ169 - 320 mg (multiple administration): 320 mg of PBTZ169 (8 capsules 40 mg) orally once per day in fasting state for 14 days
- Cohort 7: 5 healthy volunteers each of whom received a daily dose of 640 mg of PBTZ169 (16 capsules 40 mg) for 14 days
  PBTZ169 - 640 mg (multiple administration): 640 mg of PBTZ169 (16 capsules 40 mg) orally once per day in fasting state for 14 days
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Started | 6 | 6 | 6 | 6 | 6 | 5 | 5
Completed | 6 | 6 | 6 | 6 | 6 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (5.00) | 27.8 (5.64) | 31.8 (6.55) | 31.2 (6.85) | 29.0 (7.18) | 22.6 (2.61) | 28.6 (6.50) | 27.6 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 40

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Drug-related Adverse Events [Safety and Tolerability]
Description: The frequency of adverse events for which a relationship to the test drug PBTZ169 was noted
Time Frame: 14±1 days after the drug administration (up to last visit time point)
Population: Safety population: subjects who received at least one dose of PBTZ169. The population was used for the analysis and evaluation of the demographic and other baseline data and all safety parameters including AEs, physical examination, evaluation of the vital signs, previous and current therapy, ECG, all laboratory tests
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
participants | 2 | 2 | 1 | 0 | 0 | 1 | 1

2. Secondary Outcome: Peak Plasma Concentration (Сmax) of PBTZ169
Description: Up to 72 hours after the last drug administration:
  Single dosing (Cohorts 1-5): up to Day 4 (72 h after the dosing (Day 1)) Multiple dosing (Cohorts 6. 7): up to Day 17 (72 h after the last (14th) dosing)
Time Frame: Up to 72 hours after the last drug administration
Population: Pharmacokinetics analysis population (PKA): C1-5: sbjs who received PBTZ169 and had at least one measurement of PBTZ169 concentration; C6-7: sbjs who received PBTZ169 at least 7 times and had measurements of PBTZ169 concentration after the first and seventh administration.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
ng/ml
  Dosing day / Day 1 | 40.67 (15.28) | 66.99 (33.81) | 135.85 (46.32) | 156.25 (65.54) | 349.67 (145.92) | 190.82 (37.51) | 250.54 (144.33)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 243.22 (59.51) | 278.64 (70.68)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 300.55 (82.24) | 453.73 (111.85)

3. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of PBTZ169
Description: Single dosing (Cohorts 1-5): data for the dosing day (Day 1). Multiple dosing (Cohorts 6, 7): data for days 1 (1st dose), 7 and 14 (last dose)
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
h
  Dosing day / Day 1 | 2.50 [1.50 to 4.00] | 1.50 [0.75 to 3.50] | 2.00 [0.75 to 2.50] | 2.50 [0.75 to 5.00] | 1.50 [0.75 to 3.00] | 1.50 [0.50 to 4.00] | 1.50 [0.75 to 2.00]
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 2.00 [1.50 to 4.00] | 2.00 [0.75 to 4.00]
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 2.00 [1.00 to 4.00] | 2.00 [1.50 to 2.00]

4. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-∞)
Description: In the time interval from 0 to infinity
Time Frame: Up to 72 hours after the last drug administration
Population: PKA: C1-5 - SAD, C6-7 - MAD for 14 days
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
ng*h/ml
  Dosing day / Day 1 | 349.25 (206.53) | 452.83 (148.58) | 1096.36 (543.62) | 1329.65 (250.95) | 3028.04 (1286.88) | 1450.21 (586.73) | 1696.28 (993.13)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 2747.33 (795.07) | 3024.29 (726.15)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 3410.12 (1204.07) | 4358.90 (649.33)

5. Secondary Outcome: Plasma Half-life Time (T1/2) of PBTZ169
Description: as for outcome 3
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
h
  Dosing day / Day 1 | 14.306 (4.516) | 10.182 (3.663) | 16.147 (3.461) | 16.447 (2.947) | 18.175 (3.824) | 12.40 (5.72) | 9.98 (2.20)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 12.62 (5.02) | 14.16 (1.92)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 17.16 (4.35) | 17.95 (2.50)

6. Secondary Outcome: Mean Plasma Retention Time (MRT) of PBTZ169
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
h
  Dosing day / Day 1 | 15.70 (6.12) | 13.02 (4.26) | 15.44 (3.88) | 17.38 (3.68) | 19.30 (4.16) | 7.65 (0.61) | 7.70 (0.43)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 8.35 (0.75) | 8.45 (0.80)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 16.78 (1.71) | 17.89 (2.25)

7. Secondary Outcome: Total (Plasma) Clearance (Cl) of PBTZ169
Description: The Cl parameter was calculated using the following formulas: for Day 1: Cl=D/AUCinf; for Days 7 and 14: Clss=D/AUCτ
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
L/h
  Dosing day / Day 1 | 147.35 (71.97) | 190.75 (52.79) | 173.96 (69.47) | 248.08 (47.99) | 240.40 (89.12) | 244.15 (74.982) | 462.83 (197.223)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 197.223 (45.706) | 310.74 (76.273)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 146.44 (45.573) | 224.79 (42.994)

8. Secondary Outcome: Volume of Distribution (Vd) of PBTZ169
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
L
  Dosing day / Day 1 | 2762.47 (1052.08) | 2949.95 (1652.24) | 3903.25 (1354.34) | 5801.14 (1006.47) | 6359.85 (2861.493) | 3924.74 (401.074) | 6521.98 (2719.519)
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 7 |  |  |  |  |  | 2957.51 (1671.483) | 6114.55 (1680.928)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 3392.46 (2005.822) | 4067.27 (2374.585)

9. Secondary Outcome: Elimination Constant (Kel) of PBTZ169
Description: Data for doses 320 mg (Cohorts 4 and 6, total 11 volunters) & 640 mg (Cohorts 5 and 7, total 11 volunters) were combined
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
1/h | 0.052 (0.01329) | 0.077 (0.0266) | 0.063 (0.0082) | 0.066 (0.0212) | 0.066 (0.0151) | 0.066 (0.0212) | 0.066 (0.0151)

10. Secondary Outcome: Renal Clearance (Clren) of PBTZ169
Description: The renal clearance was calculated using values of the cumulative excretion in urine (from zero to 24 hours) and the area under the pharmacokinetic curve (from zero to 24 hours) (the ratio of the cumulative excretion to AUC0-24)
Time Frame: Up to 24 hours after the drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 5
mL/h
  Dosing day / Day 1 | 12.12 (7.62) | 12.64 (7.72) | 7.16 (3.80) | 11.81 (1.22) | 17.72 (6.37) | 8.5 (5.8) | 11.2 (2.9)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Day 14 |  |  |  |  |  | 5.7 (3.3) | 7.6 (3.2)

11. Secondary Outcome: Peak Steady State Plasma Concentration (Cmax,ss) of PBTZ169
Description: For cohorts 6 and 7 (multiple administration) only
Time Frame: Up to 72 hours after the last drug administration
Reporting Status: Not Posted

12. Secondary Outcome: Time to Reach Maximum Steady State Concentration (Tmax,ss) of PBTZ169
Description: For cohorts 6 and 7 (multiple administration) only
Time Frame: Up to 72 hours after the last drug administration
Reporting Status: Not Posted

13. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve in Steady State (AUCss) of PBTZ169
Description: For cohorts 6 and 7 (multiple administration) only
Time Frame: Up to 72 hours after the last drug administration
Reporting Status: Not Posted

14. Secondary Outcome: Volume of Steady State Distribution (Vd,ss) of PBTZ169
Description: For cohorts 6 and 7 (multiple administration) only
Time Frame: Up to 72 hours after the last drug administration
Reporting Status: Not Posted

15. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-t)
Description: The area under the concentration-time curve from 0 to last blood sampling
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*h/ml | 260.47 (119.06) | 381.17 (149.39) | 994.49 (462.00) | 1193.70 (212.53) | 2880.86 (1219.30)

16. Secondary Outcome: AUC0-t/AUC0-∞
Description: AUC0-t/AUC0-∞ ratio
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Number; unit: ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ratio | 0.784 | 0.829 | 0.917 | 0.899 | 0.951

ADVERSE EVENTS:
Time Frame: SAD: 14±1 days after PBTZ169 administration (Day 14±1); MAD: 21±1 days after the last (14th) PBTZ169 administration (Day 35±1).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 1/6 | 0/6 | 0/6 | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=6) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6) | Cohort 6 (N=5) | Cohort 7 (N=5)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT03036163/Prot_SAP_000.pdf